CLINICAL TRIAL: NCT02016612
Title: Seri Surgical Scaffold (TM) Support of the Lower Pole of the Breasts in Augmentation Mastopexy or Breast Reduction Patients
Brief Title: Seri Surgical Scaffold Support of the Lower Pole of the Breast
Acronym: SeriSupport
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bengtson Center (Other)
Collaborators: Allergan Medical (Industry)
Responsible Party: Principal Investigator, Bradley Bengtson, M.D., Bradley P Bengtson, MD FACS, Bengtson Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 007
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Results first posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-01

CONDITIONS: Recurrent Ptosis of the Breast
Keywords: Recurrent; Ptosis; Reduction; Mammoplasty; Mastopexy
MeSH Terms: conditions — Recurrence; Blepharoptosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Reduction, Mastopexy No Implant, No Seri (Active Comparator): Patients undergoing reduction or mastopexy but no implant is used and no Seri Surgical Scaffold support is used
  Interventions: Device: Seri Surgical Scaffold
- Mastopexy, Implant no Seri Scaffold (Active Comparator): Mastopexy with implant, No Seri Surgical Scaffold support is used
  Interventions: Device: Seri Surgical Scaffold
- Breast Reduction with Seri Support (Active Comparator): Patients undergoing breast reduction with the use of Seri Surgical scaffold support
  Interventions: Device: Seri Surgical Scaffold
- Augmentation Mastopexy, Implant and Seri (Active Comparator): Augmentation Mastopexy patients where Seri Surgical scaffold is used
  Interventions: Device: Seri Surgical Scaffold

INTERVENTIONS:
Device: Seri Surgical Scaffold — An FDA approved Bioabsorbable mesh Seri Surgical Scaffold will be utilized in the study as an internal hammock mesh support of the breast.
  Other Names: Seri; Seri Scaffold

SUMMARY:
Will the use of an FDA approved highly purified silk scaffold; Seri Surgical Scaffold help shape and hold the breast up on the chest preventing re-stretching and bottoming out of the breast in breast reduction or augmentation-mastopexy patients? The amount of stretch will be measured manually as well as percent of breast tissue measured with the Canfield Vectra 3-D Imaging system reporting the amount of breast tissue above and below the nipple level.

DETAILED DESCRIPTION:
Patients having augmentation mastopexy or breast reduction will be informed about Seri Scaffold and allowed to have Seri support included in their surgery or not. If the choose the scaffold will be placed under the skin in the lower pole of the breast as an internal hammock to help take weight off of the breast and potentially help prevent future stretch of the lower pole.

ELIGIBILITY:
Inclusion Criteria:

Age =>18 years

* requesting procedure
* No active cancer or infection

Exclusion Criteria:

* Known allergy to silk
* Pregnant or lactating

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-10; Primary Completion 2015-11 (Actual); Study Completion 2016-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley P Bengtson, MD, Principal Investigator — Bengtson Center
Locations (2):
- United States (2):
  - Bengtson Center for Aesthetics and Plastic Surgery, Grand Rapids, Michigan
  - Center for Aesthetics and Plastic Surgery, Grand Rapids, Michigan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Reduction, Mastopexy No Implant, No Seri: Patients undergoing reduction or mastopexy but no implant is used and no Seri support
  Seri Surgical Scaffold: An FDA approved Bioabsorbable mesh Seri Surgical Scaffold will be utilized in the study as an internal hammock mesh support of the breast.
- Mastopexy, Implant no Seri Scaffold: Mastopexy with implant, No Seri support is used
  Seri Surgical Scaffold: An FDA approved Bioabsorbable mesh Seri Surgical Scaffold will be utilized in the study as an internal hammock mesh support of the breast.
- Breast Reduction With Seri Support: Patients undergoing breast reduction with the use of Seri support
  Seri Surgical Scaffold: An FDA approved Bioabsorbable mesh Seri Surgical Scaffold will be utilized in the study as an internal hammock mesh support of the breast.
- Augmentation Mastopexy, Implant and Seri: Augmentation Mastopexy patients where Seri Scaffold is placed
  Seri Surgical Scaffold: An FDA approved Bioabsorbable mesh Seri Surgical Scaffold will be utilized in the study as an internal hammock mesh support of the breast.
Period: Overall Study
Arm/Group | Reduction, Mastopexy No Implant, No Seri | Mastopexy, Implant no Seri Scaffold | Breast Reduction With Seri Support | Augmentation Mastopexy, Implant and Seri
Started | 25 | 25 | 26 | 61
Completed | 25 | 25 | 26 | 61
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reduction, Mastopexy No Implant, No Seri | Mastopexy, Implant no Seri Scaffold | Breast Reduction With Seri Support | Augmentation Mastopexy, Implant and Seri | Total
Number analyzed (Participants) | 25 | 25 | 26 | 61 | 137
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 26 | 61 | 137
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 47 [20 to 63] | 38 [20 to 56] | 48 [39 to 65] | 37 [26 to 65] | 42 [20 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 26 | 61 | 137
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 3 | 0 | 5
  White | 22 | 23 | 22 | 61 | 128
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 25 | 26 | 61 | 137

OUTCOME MEASURES:

1. Primary Outcome: Nipple to Fold Measurement on Stretch
Description: The Nipple to fold will be measured manually over time to 1 year
Time Frame: 1 year post op
Measure: Mean (Full Range); unit: centimeters
Arm/Group | Reduction, Mastopexy No Implant, No Seri | Mastopexy, Implant no Seri Scaffold | Breast Reduction With Seri Support | Augmentation Mastopexy, Implant and Seri
Number analyzed (Participants) | 25 | 25 | 26 | 61
centimeters | 2.3 [1.2 to 4.2] | 2.5 [1.2 to 4.1] | 1.4 [0.5 to 2.6] | 1.4 [0.7 to 2.6]

2. Secondary Outcome: Percent Breast Tissue Above Nipple
Description: The percentage of breast tissue above and below the horizontal plane of the nipple over time
Time Frame: 1 year post op
Measure: Mean (Full Range); unit: percentage of volume
Arm/Group | Reduction, Mastopexy No Implant, No Seri | Mastopexy, Implant no Seri Scaffold | Breast Reduction With Seri Support | Augmentation Mastopexy, Implant and Seri
Number analyzed (Participants) | 25 | 25 | 26 | 61
percentage of volume | 35 [0.0 to 100] | 30 [0 to 100] | 15 [0 to 100] | 18 [0 to 100]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Reduction, Mastopexy No Implant, No Seri | Mastopexy, Implant no Seri Scaffold | Breast Reduction With Seri Support | Augmentation Mastopexy, Implant and Seri
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 3/26 | 2/61
Other Adverse Events (participants affected / at risk) | 3/25 | 2/25 | 3/26 | 2/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reduction, Mastopexy No Implant, No Seri (N=25) | Mastopexy, Implant no Seri Scaffold (N=25) | Breast Reduction With Seri Support (N=26) | Augmentation Mastopexy, Implant and Seri (N=61)
seroma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2) — seroma and partial Seri removal
dehiscence (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2) — skin dehiscence
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reduction, Mastopexy No Implant, No Seri (N=25) | Mastopexy, Implant no Seri Scaffold (N=25) | Breast Reduction With Seri Support (N=26) | Augmentation Mastopexy, Implant and Seri (N=61)
skin dehiscence (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 3 (3) | 2 (2) — skin dehiscence
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Superficial infection limited to the skin

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No